CLINICAL TRIAL: NCT03606473
Title: Exploration of Mechanisms of Effects of Prenatal Cocaine Exposure in Young Adults
Brief Title: Brain Mechanisms in Young Adults
Acronym: MHP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gale Richardson (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Gale Richardson, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO17080203
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Cocaine-Related Disorders
Keywords: prenatal exposure
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Dextroamphetamine

STUDY DESIGN:
Intervention Model Description: [C-11]NPA d-amphetamine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prenatal cocaine exposed subjects (Experimental): [C-11]NPA PET at baseline and post d-amphetamine
  Interventions: Drug: d-amphetamine; Radiation: [C-11]NPA
- Comparison subjects (Experimental): [C-11]NPA PET at baseline and post d-amphetamine
  Interventions: Drug: d-amphetamine; Radiation: [C-11]NPA

INTERVENTIONS:
Drug: d-amphetamine — is used to stimulate dopamine release in the brain
Radiation: [C-11]NPA — PET radiotracer

SUMMARY:
The goal of this study is to use [C-11]NPA and amphetamine (oral, 0.5 mg/kg) to measure striatal dopamine transmission in prenatal cocaine exposed subjects (PCE) and comparison subjects (COMP)

DETAILED DESCRIPTION:
Prenatal cocaine exposure (PCE) has consistently been associated with behavioral deficits through childhood, adolescence, and young adulthood in our ongoing study (PRO15080516 - Effects of Prenatal Cocaine Use: 25-Year Follow-Up). Further, 21-year-olds with PCE in our study were twice as likely to have been arrested as non-exposed offspring, were more likely to be diagnosed with Conduct Disorder, had higher disinhibition scores, were significantly more likely to use alcohol and marijuana earlier, and to have earlier sexual intercourse. The effects of PCE on the developing nervous system may cause changes in brain function that underlie these behavioral outcomes.

This study seeks to examine dopamine (DA) transmission in vivo, using positron emission tomography (PET) with [C-11]NPA, in striatal regions of interest in subjects who have a history of exposure to prenatal cocaine (PCE). We hypothesize that PCE is associated with increases in dopamine in the striatum relative to COMP. This may explain the impulsivity and high risk behaviors in PCE subjects

ELIGIBILITY:
All potential subjects are current participants in the larger parent study entitled "Effects of Prenatal Cocaine Exposure: 25-Year Follow-Up", IRB PRO15080516. Participants are between 25 and 30 years of age.

Inclusion Criteria:

* Prenatal cocaine exposed subjects (PCE): Offspring exposed to prenatal cocaine (concurrent exposure to prenatal alcohol and tobacco are not exclusionary) as determined by detailed interviewing during pregnancy
* Comparison group (COMP): Offspring NOT exposed to prenatal cocaine (exposure to prenatal alcohol and tobacco are not exclusionary) as determined by detailed interviewing during pregnancy.

Exclusion criteria for both PCE and COMP groups:

* No current mania or psychosis based on current mental status exam and SCID-IV modules A (pages A18-A37) and B (pages B1-B8);
* No current cocaine, heroin, opioid, methadone, benzodiazepine, methamphetamine use (negative urine drug screen at both day of screening and the day of PET scan);
* No current use of cannabis (a negative urine drug screen on day of PET scan; Note: a positive cannabis urine on the day of screening will not be exclusionary because cannabis tends to be used for recreation; and it takes a long time for it turn negative because it is released from fat cells in body long after subject has quit; and it has been shown to not impact amphetamine-induced dopamine release in prior studies);
* Not currently taking prescription or over the counter medications that can alter monoamine transmission in the brain or interact with the d-amphetamine challenge or alter amphetamine concentrations (major CYP2D6 inhibitors such as fluoxetine, thioridazine, terbinafine etc., as well as pseudo-ephedrine, atomoxetine, SSRIs, etc.);
* No use of acidifying (fruit juice; beverages; ascorbic acid) and alkalinizing agents (such as sodium bicarbonate) that alter amphetamine concentrations at least 12 hrs before PET scan day;
* No current or past severe medical or neurological illnesses such as seizure disorders, head injury with prolonged loss of consciousness, hypertension, prior MI, CAD etc., (determined by physician investigator's elicited medical history, physical exam, review of labs, and EKG results);
* Not currently pregnant (serum pregnancy test at screening) or breastfeeding;
* No history of radioactivity exposure via prior nuclear medicine studies or occupational exposure in past 12 months;
* No metallic objects in the body that are contraindicated for MRI;
* SBP > 135, DBP > 85, and/or HR ≤ 50 or ≥ 100 (documented before the PET scans; Note: it is not unusual to have to repeat screening vital signs in subjects' because some subjects tend to have white coat syndrome and present with elevated vitals at screening, which later normalizes);
* No first-degree relative with an MI or stroke or TIA prior to 50 years of age;
* No first-degree relative with psychosis or mania.

Ages: 25 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Percent change in Binding potential (BPnd) | Baseline BPnd (time 0) and Post-amphetamine BPnd (time 3 hours
  DELTA BPND

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No